CLINICAL TRIAL: NCT03971019
Title: Survival Benefits of Statins in Breast Cancer Patients With Abnormal Lipid Metabolism
Brief Title: Survival Benefits of Statins in Breast Cancer Patients
Acronym: SBSBC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-SBSBC
Record Dates: First submitted 2019-03-30; First posted 2019-06-03 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; statins; abnormal lipid metabolism
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Control Groups; Diet

STUDY DESIGN:
Intervention Model Description: A randomized, open, blank controlled, single-center clinical trial. The control group used dietary intervention instead of statins.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin therapy (experimental group) (Experimental): On the basis of guiding patients to control their diet and improve their lifestyle, etc.
  Simvastatin 20mg/d QN Po (dosage can be adjusted according to the blood lipid level of each reexamination) Atorvastatin 10mg/d QN Po (patients who cannot tolerate the side effects of simvastatin may consider replacing this drug)
  Interventions: Drug: statins
- Dietary intervention group (control group) (Other): Guiding patients to control diet, improve lifestyle, etc.
  Interventions: Behavioral: Dietary intervention group (control group)

INTERVENTIONS:
Drug: statins — On the basis of dietary intervention. Simvastatin 20mg/d QN Po (half an hour before bedtime) (dosage can be adjusted according to other indicators of blood lipid level in each review), atorvastatin 10mg/d QN Po (half an hour before bedtime) (patients who can not tolerate the side effects of simvastatin can consider replacing this drug).
  Other Names: Simvastatin Shu Jiangzhi is manufactured by Merchant Company20mg*14 tablets Dose group: 20 mg once a day before bed; Atorvastatin Lipitor, commonly known as Atorvastatin Calcium Tablets, 20mg*7 tablets Dose group: 10 mg once a day before bed; Atorvastatin Ale Beijing Jialin Pharmaceutical Co., Ltd. Alatorvastatin Calcium Tablets Specification and packing: 10mg*7 tablets Dose group: 10 mg once a day before bed
  Arms: Statin therapy (experimental group)
Behavioral: Dietary intervention group (control group) — Restriction of dietary components that increase LDL-C Saturated Fatty Acids Less than 7% of total energy Dietary cholesterol < 300 mg/d Increasing Dietary Ingredients for Reducing LDL-C Phytosterol 2~3 g/d Water soluble dietary fiber 10~25 g/d total energy Adjusted to maintain ideal weight or lose weight Physical activity Maintain moderate intensity exercise and consume at least 200 kcal of calories per day
  Other Names: Dietary and motor regulation
  Arms: Dietary intervention group (control group)

SUMMARY:
In this study, we compared the survival benefit of breast cancer patients with dyslipidemia (low and medium risk of ASCVD). The control group used dietary intervention instead of statins intervention. The main endpoint was 5 years DFS. The subjects were breast cancer patients.

DETAILED DESCRIPTION:
A randomized, open, blank controlled, single-center clinical trial was conducted to compare the survival benefits of statins in breast cancer patients with dyslipidemia (low and medium risk of ASCVD). The control group used dietary intervention instead of statins. The main endpoint was 3 and 5 years DFS. The subjects were breast cancer patients. In this study, 348 patients were randomly divided into two groups according to patients' wishes and written informed consent. The experimental group: control group = 1:1. Subjects were screened and administered continuously until the disease progressed and the toxicity was intolerable. Informed consent was withdrawn or the researcher decided that the drug must be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as invasive breast cancer, it has been treated surgically, confirmed by histology, cytology or imaging.
2. Female patients (35-75 years old);
3. The low-risk patients with ASCVD are detailed in Annex 1.
4. Signed written informed consent approved by IRB or IEC

Exclusion Criteria:

1. The subjects were pregnant or lactating.
2. Pregnancy test positive (urine or serum) in women with potential pregnancy within 7 days before administration.
3. Other invasive tumors (including the second primary breast cancer) may affect the evaluation of outcomes and the compliance of schemes, but subjects who have been cured and survived disease-free for at least five years can be selected.
4. Patients with chronic underlying liver diseases who have abnormal liver function and/or clinical manifestations:

   Serum total bilirubin > 2.5 *ULN; or INR > 1.5 although there was no increase in bilirubin Serum ALT or AST > 3 *ULN; Alkaline phosphatase > 2.5 *ULN; Elevated ALT or AST may gradually recover, but with progressively increased fatigue, nausea and vomiting, fever, right upper abdominal pain or tenderness.
5. Extremely high risk ASCVD patients Including acute coronary syndrome (ACS), stable coronary heart disease, revascularization, ischemic cardiomyopathy, ischemic stroke, transient ischemic attack, peripheral atherosclerosis, etc.
6. High-risk ASCVD patients (in accordance with one of the following circumstances):

   LDL-C>4.9 mmol/L or TC>7.2 mmol/L Diabetic patients with 1.8 mmol/L < LDL-C < 4.9 mmol/L (or) 3.1 mmol/L < TC < 7.2 mmol/L and age < 40 years

   The 10-year risk of ASCVD was moderate and younger than 55 years old. The remaining life risk was assessed. Those with any of the following two or more risk factors are defined as high risk:

   Systolic or diastolic blood pressure (> 160 mmHg) or (> 100 mmHg)
   * Non-HDL-C>5.2 mmol/L (200 mg/dl)
   * HDL-C < 1.0 mmol/L (40 mg/dl)
   * BMI>28 kg/m2 Smoking
7. In the abnormal group of simple TG (triglyceride), TG (> 5.7 mmol/L)
8. Other serious diseases, including:

   Congestive heart failure (NYHA grade II, III, IV); dyspnea at rest or requiring oxygen therapy; severe infection; uncontrolled diabetes mellitus;
9. If there are serious mental or mental disorders, it is estimated that the subjects'compliance to participate in this study is not strong.
10. Drug allergies to research drugs are known.
11. Participated in other drug clinical trials in the past 30 days.
12. Failure to complete at least one cycle of clinical trials based on this protocol, and failure to evaluate safety and effectiveness.
13. Serious violation of this study program, not in accordance with the prescribed dose, method and course of treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer patients
Enrollment: 314 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 years
  Disease free survival

SECONDARY OUTCOMES:
OS | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, M.D., Principal Investigator — PUMCH
Locations (1):
- PUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The results of this study can be shared

REFERENCES:
- [Background] Filippatos TD, Liberopoulos EN, Pavlidis N, Elisaf MS, Mikhailidis DP. Effects of hormonal treatment on lipids in patients with cancer. Cancer Treat Rev. 2009 Apr;35(2):175-84. doi: 10.1016/j.ctrv.2008.09.007. Epub 2008 Nov 14. PMID 19013720
- [Result] Patnaik JL, Byers T, DiGuiseppi C, Dabelea D, Denberg TD. Cardiovascular disease competes with breast cancer as the leading cause of death for older females diagnosed with breast cancer: a retrospective cohort study. Breast Cancer Res. 2011 Jun 20;13(3):R64. doi: 10.1186/bcr2901. PMID 21689398
- [Result] Beckwitt CH, Brufsky A, Oltvai ZN, Wells A. Statin drugs to reduce breast cancer recurrence and mortality. Breast Cancer Res. 2018 Nov 20;20(1):144. doi: 10.1186/s13058-018-1066-z. PMID 30458856
- [Result] Liu B, Yi Z, Guan X, Zeng YX, Ma F. The relationship between statins and breast cancer prognosis varies by statin type and exposure time: a meta-analysis. Breast Cancer Res Treat. 2017 Jul;164(1):1-11. doi: 10.1007/s10549-017-4246-0. Epub 2017 Apr 21. PMID 28432513

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03971019/Prot_SAP_ICF_001.pdf